CLINICAL TRIAL: NCT02283463
Title: Patient Discomfort With a Novel Suction Based Cervical Retractor Compared to the Traditional Cervical Tenaculum
Brief Title: Novel Cervical Retraction Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioceptive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AB001
Record Dates: First submitted 2014-10-30; First posted 2014-11-05 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Pain Due to Certain Specified Procedures
MeSH Terms: interventions — Intrauterine Devices; Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Standard Cervical Tenaculum (Active Comparator): Single tooth tenaculum, pierces the tissue of the cervix to allow provider to stabilize and place traction on the cervical cal/uterus
  Interventions: Device: Intrauterine device (IUD) insertion; Procedure: Endometrial biopsy
- Bioceptive Cervical Retraction Device (Experimental): Suction based method for stabilizing the cervix and uterus. Achieves suction 360 degrees around cervical os creating a portal through which instruments can be passed into the cervical canal and uterus. Provider can still place traction on uterus with this device just as with tenaculum.
  Interventions: Device: Intrauterine device (IUD) insertion; Procedure: Endometrial biopsy

INTERVENTIONS:
Device: Intrauterine device (IUD) insertion
Procedure: Endometrial biopsy

SUMMARY:
This study will test a suction-based method of engaging the cervix. Bioceptive has developed a device that more gently and atraumatically attaches to the cervix with no bleeding. This novel attachment mechanism may diminish pain and discomfort. Pre-clinical testing has been performed on the device including testing on synthetic uterine models, human cadavers, and human uteri immediately post-hysterectomy (Utah IRB # 00059096). Results from these efforts have shown effective attachment to the cervix and the ability for the device to maintain suction throughout a procedure atraumatically. This study proposes to introduce this minimal risk device in a clinical setting to determine the response of women undergoing gynecologic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting for IUD insertion or endometrial biopsy
* Able to consent for study in English or Spanish

Exclusion Criteria:

* Post-menopausal
* Current pregnancy
* Cervical abnormalities (cervical polyp, cervical lesion, or irregularity)
* Use of narcotics or Benzodiazepines prior to procedure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-09; Primary Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measure 100 point visual analogue scale | 1 day
  Pain recorded by patient during the procedure and one day following via 100 point visual analogue scale. (0 = none, 100 = worst imaginable)

SECONDARY OUTCOMES:
Procedural Satisfaction Patient records level of satisfaction with the procedure (Very Unsatisfied, Unsatisfied, Neutral, Satisfied, Very Satisfied) | < 1 hour
  Patient records level of satisfaction with the procedure (Very Unsatisfied, Unsatisfied, Neutral, Satisfied, Very Satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, MPH, Principal Investigator — University of Utah, Dept. of Obstetrics and Gynecology
Locations (1):
- University of Utah, School of Medicine, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Turok DK, Simmons RG, Cappiello B, Gawron LM, Saviers-Steiger J, Sanders JN. Use of a novel suction cervical retractor for intrauterine device insertion: a pilot feasibility trial. BMJ Sex Reprod Health. 2018 Nov 5:bmjsrh-2017-200031. doi: 10.1136/bmjsrh-2017-200031. Online ahead of print. PMID 30396906